CLINICAL TRIAL: NCT07378566
Title: Digitally Supported Intervention to Master Complex Fall Risk Situations in Persons With Multiple Sclerosis - a Multicenter Study (STAR)
Brief Title: Intervention to Master Complex Fall Risk Situations in Persons With Multiple Sclerosis (STAR)
Acronym: STAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Institution of Medical Sciences, Örebro University (Unknown); Region Gävleborg (Other); Region Västmanland (Other); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Ylva Nilsagard, Research leader Integrated care, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 285079
Record Dates: First submitted 2025-09-03; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Fall
Keywords: falls; prevention
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two phases starting with an internal pilot study followed by a full scale RCT
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This arm will receive an individual analyses of current fall situations and a tailored individual strategy aiming to reduce fall frequency
  Interventions: Behavioral: Individual strategies
- Control group (No Intervention): This arm will only receive general advice. Will be offered the intervention after ending of the study period

INTERVENTIONS:
Behavioral: Individual strategies — This arm will receive an individual analyses of current fall situations and a tailored individual strategy aiming to reduce fall frequency
  Arms: Intervention group

SUMMARY:
People with multiple sclerosis (MS) have a higher fall risk compared to older people and to the general population. A meta-analysis reported that 56% of those with mild to moderate MS, fell at least once during a 3-month period. The risk of falling seems to peak when the walking distance starts to be affected and when walking aids are introduced and the walking distance is as short as 100 m. Previous studies have identified a number of fall risk factors, both relating to MS- symptoms and contextual factors. In a study published in 2025, we reported the complexity of fallsituations and the interaction between triggering factors, contextual factors and activities and circumstances that occurred before the fall incidents . The symptoms when having MS varies between individuals as well as over time. I the planned randomised, controlled multicenter study we move forward, producing individual fallrisk analyses based upon the findings from the study published in 2025, and offer individual strategies. This has not been studied before. All participants will receive general information on how fall risk can be prevented. Those randomised to control group will be offered the intervention after ending of the study. The study will be conducted in two phases starting with an internal pilot study followed by a full scale randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The intervention will be based on previous findings i. e., fall risk factors related to the International Classification of Functioning, Disability and Health and is an add-on intervention to a general fall risk information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS
* Affected ability to walk du to MS according to the participant
* At least one self-reported fall the last 3 months due to MS according to the participant

Exclusion Criteria:

* Unable to walk 100m even with walking device and/or pauses.
* Apparently affected walking ability due to other conditions such as for example orthopedic or other neurological diseases.
* Difficulty to answer questionnaires written in Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prospectively self-reported falls (rate, time to fall) | every 14th day during 6 months
  Self-reported falls collected every two weeks during a 6-month period

SECONDARY OUTCOMES:
Falls-Efficacy Scale-International score | baseline and immediately after the intervention
  16 questions regarding level of concern about falling. Scores for each item together adds up to a total that ranges as follows: 16 (no concerns about falling( to 28 (severe concern about falling
Activity-specific balance Confidence Scale score | baseline and immediately after the intervention
  16 questions regarding confidence to remain balance during everyday activities scoring from 0 (no confidence) to 100 (full confidence)
Self-rated ability to reduce falls | baseline and immediately after the intervention
  One question measured using a visual analogue scale 0 (no ability) to 100 (full ability)
Self-rated ability to understand one's own fall risk factors | baseline and immediately after the intervention
  One question using a visual analogue scale 0 (no understanding) to 100 (full understanding)
Self-rated fear of falling reducing activities | baseline and immediately after the intervention
  One question where the person rates whether fear of falling have made them do less activities compared to before (yes, no, don't know, prefer not to answer)
12-item MS Walking scale score | baseline and immediately after the intervention
  Measures self-rated affected walking ability due to MS using 12 items. A score is obtained by subtracting the minimum score possible (=12) from the achieved sum, dividing by the range (=48) and multiplying by 100. Higher scores indicate more limited walking ability

OTHER OUTCOMES:
Timed Up and Go test | baseline
  Measures basic mobility (time for rising up from a chair, walk 3m, turn around, walk back and sit down.
Six Spot Step Test | baseline
  Measures speed, coordination and balance using time for a person to walk in zic-zac, kicking bricks using one foot for round one and the other foot for round two.
Symbol Digit Modalities Test | baseline
  Screening test for cognitive function pairing geometric figures with 10 numbers. Number of right and wrong answers given during 90 seconds
"Frändin Grimby" activity scale | baseline and immediately after the intervention
  Measures physical activity the past 6 months using six alternatives ranging from hardly no physical activity to very hard physical activity
MS Impact Scale-29 | baseline
  Measures self-rated physical and psychological MS-specific outcomes the past two weeks ranging from not at all to extremely. summing responses for its 20-item Physical Scale and 9-item Psychological Scale. The raw scores are transformed to a 0-100 scale, where higher scores indicate greater impact from the disease. The transformation for the Physical Scale is (100*(observed score - 20)) / (100-20), and for the Psychological Scale is (100*(observed score - 9)) / (45-9). A responder specific mean score can be calculated from completed items if at least 50% of the items in a scale are answered.

CONTACTS AND LOCATIONS:
Overall Officials: Ylva E Nilsagård, Ass. prof, Principal Investigator — University Healthcare Research Center, Faculty of Medicine and Health

IPD SHARING:
Plan to Share IPD: Yes
We aim to publish a study protocol that includes a full description of the study
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and Statistical Analysis plan before study start.
Access Criteria: Open access if accepted for publication

REFERENCES:
- [Result] Salari N, Darvishi N, Ahmadipanah M, Shohaimi S, Mohammadi M. Global prevalence of falls in the older adults: a comprehensive systematic review and meta-analysis. J Orthop Surg Res. 2022 Jun 28;17(1):334. doi: 10.1186/s13018-022-03222-1. PMID 35765037
- [Result] Mazumder R, Murchison C, Bourdette D, Cameron M. Falls in people with multiple sclerosis compared with falls in healthy controls. PLoS One. 2014 Sep 25;9(9):e107620. doi: 10.1371/journal.pone.0107620. eCollection 2014. PMID 25254633
- [Result] Nilsagard Y, Gunn H, Freeman J, Hoang P, Lord S, Mazumder R, Cameron M. Falls in people with MS--an individual data meta-analysis from studies from Australia, Sweden, United Kingdom and the United States. Mult Scler. 2015 Jan;21(1):92-100. doi: 10.1177/1352458514538884. Epub 2014 Jun 16. PMID 24948687
- [Result] Gunn HJ, Newell P, Haas B, Marsden JF, Freeman JA. Identification of risk factors for falls in multiple sclerosis: a systematic review and meta-analysis. Phys Ther. 2013 Apr;93(4):504-13. doi: 10.2522/ptj.20120231. Epub 2012 Dec 13. PMID 23237970
- [Result] Carling A, Forsberg A, Nilsagard Y. Falls in people with multiple sclerosis: experiences of 115 fall situations. Clin Rehabil. 2018 Apr;32(4):526-535. doi: 10.1177/0269215517730597. Epub 2017 Sep 13. PMID 28901164
- [Result] Nilsagard Y, Lundholm C, Denison E, Gunnarsson LG. Predicting accidental falls in people with multiple sclerosis -- a longitudinal study. Clin Rehabil. 2009 Mar;23(3):259-69. doi: 10.1177/0269215508095087. PMID 19218300
- [Result] Gunn H, Creanor S, Haas B, Marsden J, Freeman J. Risk factors for falls in multiple sclerosis: an observational study. Mult Scler. 2013 Dec;19(14):1913-22. doi: 10.1177/1352458513488233. Epub 2013 Apr 30. PMID 23633067
- [Result] Waneskog AH, Forsberg AS, Nilsagard YE. Exploring the Complexity of Falls in People With Multiple Sclerosis: A Qualitative Study. Int J MS Care. 2024 Nov 5;26(Q4):308-314. doi: 10.7224/1537-2073.2024-020. eCollection 2024 Oct. PMID 39502367

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT07378566/Prot_SAP_000.pdf